CLINICAL TRIAL: NCT06121635
Title: The Effects of Transcranial Direct Current Stimulation and Transcutaneous Spinal Direct Current Stimulation on Robot-assisted Gait Training in Patients With Multiple Sclerosis
Brief Title: The Effects of Two Types of t-DCS Stimulation on Robot-assisted Gait Training in Patients With Multiple Sclerosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Gulser CINBAZ, research assistant, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09.2020.1075
Record Dates: First submitted 2023-10-23; First posted 2023-11-08 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Multiple Sclerosis; Transcranial Direct Current Stimulation
MeSH Terms: conditions — Multiple Sclerosis | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Participants will not be informed whether the stimulations applied are active or sham.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ts-DCS Group (Experimental): Active ts-DCS and sham t-DCS will be applied simultaneously. 2mA intensity ts-DCS will be applied, with the active electrode being the cathode. The cathode will be placed the spinous process of T10 vertebral process, while the anode will be placed on the left deltoid. 2mA intensity t-DCS will be applied, with the active electrode being the anode. The International EEG 10/20 System will be used to electrode placement. The anode will be placed on the left M1, while the catode will be placed on the right supraorbital region. In the sham application, the placement of the electrodes will be the same as the active stimulation but It's will be stopped after 30 seconds. This sham procedure has been reported to be a good pseudostimulation method. ts-DCS and t-DCS will be administered using a stimulator (TCT Research Limited, Hong Kong). In both stimulations, 2 electrodes (35 cm2) immersed in saline solution will be used. The stimulations will be applied in 20 min sessions, 3 days/4 weeks.
  Interventions: Combination Product: Transcutaneous Spinal Direct Current Stimulation and Transcranial Direct Current Stimulation
- t-DCS Group (Experimental): Active t-DCS and sham ts-DCS will be applied simultaneously. 2mA intensity t-DCS will be applied, with the active electrode being the anode. The International EEG 10/20 System will be used to electrode placement. The anode will be placed on the left M1, while the catode will be placed on the right supraorbital region. 2mA intensity ts-DCS will be applied, with the active electrode being the cathode. The cathode will be placed the spinous process of T10 vertebral process, while the anode will be placed on the left deltoid. In the sham application, the placement of the electrodes will be the same as the active stimulation but It's will be stopped after 30 seconds. This sham procedure has been reported to be a good pseudostimulation method. ts-DCS and t-DCS will be administered using a stimulator (TCT Research Limited, Hong Kong). In both stimulations, 2 electrodes (35 cm2) immersed in saline solution will be used. The stimulations will be applied in 20 min sessions, 3 days/4 weeks.
  Interventions: Combination Product: Transcutaneous Spinal Direct Current Stimulation and Transcranial Direct Current Stimulation
- Control Group (Sham Comparator): Sham ts-DCS and sham t-DCS will be applied simultaneously. 2mA intensity ts-DCS will be applied, with the active electrode being the cathode. The cathode will be placed the spinous process of T10 vertebral process, while the anode will be placed on the left deltoid. 2mA intensity t-DCS will be applied, with the active electrode being the anode. The International EEG 10/20 System will be used to electrode placement. The anode will be placed on the left M1, while the catode will be placed on the right supraorbital region. In both stimulations, the placement of the electrodes in Sham application will be the same as in active stimulation, but it will be stopped after 30 seconds. ts-DCS and t-DCS will be administered using a stimulator (TCT Research Limited, Hong Kong). In both stimulations, 2 electrodes (35 cm2) immersed in saline solution will be used. The stimulations will be applied in 20 min sessions, 3 days/4 weeks.
  Interventions: Combination Product: Sham ts-DCS and sham t-DCS

INTERVENTIONS:
Combination Product: Transcutaneous Spinal Direct Current Stimulation and Transcranial Direct Current Stimulation — At the robot-assisted gait training, 20-minute gait training for the patient at an appropriate speed with the Locohelp Woodway device. The aim is to re-teach proper walking, gait cycle timing, and create a near-normal gait pattern through multiple repetitions. Robot-assisted gait training will be performed immediately following the stimulation applied to the patients.
  Other Names: robot-assisted gait training
  Arms: t-DCS Group; ts-DCS Group
Combination Product: Sham ts-DCS and sham t-DCS — Sham ts-DCS and sham t-DCS
  Arms: Control Group

SUMMARY:
The primary aim of this study is to determine the transcranial direct current stimulation and transcutaneous spinal direct current stimulation in addition to robot-assisted walking training in individuals with Multiple sclerosis; to examine the effects on motor functions against each other and sham application. Secondary aim of this study is to show the relation of these effects with tDCS and ts-DCS through fatigue and quality of life evaluations.

DETAILED DESCRIPTION:
These study is planned to be carried out in the Cadde Medical Center clinic. The patients who will participate in the study will be determined according to the inclusion criteria among the patients who applied to the Multiple Sclerosis Outpatient Clinic of Istanbul Medeniyet University Göztepe Research Hospital, Department of Neurology. As a result of the power analysis, 36 participants were planned to be included in the study. 20 minutes of non-invasive brain stimulation will be applied to the individuals participating in these study before the 20 minutes robot-assisted walking training (RATG), 3 days a week for 4 weeks. Participants will be divided into 3 groups according to the type of stimulation applied by simple randomization. These groups are 1) anodal tDCS + sham ts-DCS; 2) sham tDCS + cathodal ts-DCS 3) sham tDCS + sham ts-DCS. The same evaluations will be applied to all participants during the study and the evaluations are planned as before and after the intervention. The data collected as a result of the evaluations will be analyzed with SPSS version 22.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with MS and suffering from walking difficulties due to MS
* EDSS score between 2-6
* Being over 18 years old

Exclusion Criteria:

* Relapsed within the last two months
* Changed medication within 45 days
* Hospitalized in the last three months
* Had other neurological or musculoskeletal problems
* Had an obstacle to stimulation (skin problems, metal implants, etc.)
* Do not want to participate in the study individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Timed 25-Foot Walk (T25-FW) | 4 weeks
  Timed 25 Foot Walking Test was used for objective evaluation of walking. In T25-FW, which evaluates lower extremity function, the individual is asked to walk 25 steps as quickly and safely as possible (if he/she uses a walking aid, this is done together). The time spent walking is recorded in seconds.
Time Up and Go (TUG) | 4 weeks
  It is a performance-based test used to evaluate functional mobility and walking speed. The person is asked to get up from the chair he/she is sitting on without support from his/her arms, walk 3 meters at a safe and normal speed, turn around, walk back, sit on the chair again, and the time is recorded in seconds (sec). The test is started with the patient's feet flat on the floor and arms resting on the armrest of the chair. Three repetitions are made and the best result is recorded.
Multiple Sclerosis Walking Scale-12 (MSWS-12) | 4 weeks
  It is a 12-item rating scale used to assess individuals' perspectives on the impact of their disease on their ability to walk. During the test, patients are asked to rate how much MS affects their mobility, such as standing, walking, running, and climbing stairs, on a 5-point Likert Scale (1=almost not at all, 5=extremely). A high score indicates that walking ability is affected or the patient has difficulty walking. The lowest score can be 12 and the highest score can be 60 from the test.
Gait Speed Assessment | 4 weeks
  Calculation of walking speed will be done by 2D video analysis method. Kinovea 2D motion analysis software (GPLv2 license, 2019) will be used for analysis. The method has validity and reliability. The videos taken with the cameras placed laterally will be uploaded to the program and the necessary calculations will be made.

SECONDARY OUTCOMES:
Fatigue Severity Scale (FSS) | 4 weeks
  The scale, which includes the experience of fatigue, its causes and its effects on daily life, consists of 9 questions and is a Likert-type scale where each question takes a value between 0 and 7. The highest score reached is 63. A score of 36 or above indicates a high perception of fatigue severity.
Fatigue Impact Scale (FIS) | 4 weeks
  FIS will be used to evaluate the reflection of fatigue on daily activities in patients. This scale evaluates the physical, cognitive and social effects of fatigue in the last month with a total of 40 questions (0 = no problem, 4 = extreme). The total score ranges from 0-160, with higher scores indicating a higher degree of fatigue impact

CONTACTS AND LOCATIONS:
Locations (1):
- Cadde Tıp Merkezi, Istanbul, Kadıköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No